CLINICAL TRIAL: NCT03817060
Title: CuMulativE Live bIrth Rate of Patients at High Risk of OHSS After Freeze-all Embryos at Cleavage or blAstocyst Stage in a Single Embryo Transfer Setting (MELISSA)
Brief Title: CuMulativE Live bIrth Rate of Patients at High Risk of OHSS After Freeze-all Embryos at Cleavage or blAstocyst Stage
Acronym: MELISSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Theoni Tarlatzi, Principal Investigator, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRB_201807_150
Record Dates: First submitted 2018-12-07; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Infertility
Keywords: OHSS; Agonist trigger; freeze-all; blastocyst; cleavage
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cleavage (Active Comparator): Embryos cryopreserved with vitrification at the cleavage stage (day 3) of embryo development
  Interventions: Procedure: cryopreservation of embryos at cleavage stage
- Blastocyst (Active Comparator): Embryos cryopreserved with vitrification at the blastocyst stage (day 5 or 6)
  Interventions: Procedure: cryopreservation of embryos at blastocyst stage

INTERVENTIONS:
Procedure: cryopreservation of embryos at cleavage stage — cryopreservation of embryos at cleavage stage (day 3) of embryo development
  Arms: Cleavage
Procedure: cryopreservation of embryos at blastocyst stage — cryopreservation of embryos at blastocyst stage (day 5 or 6) of embryo development
  Arms: Blastocyst

SUMMARY:
Ovarian stimulation for the induction of multifollicular growth by gonadotrophins represents an important part of In Vitro Fertilization (IVF). However, the use of these drugs can be associated with side effects, from which the most common is the Ovarian Hyperstimulation Syndrome (OHSS). Stimulation with gonadotrophins in a Gonadotropin-releasing hormone (GnRH) antagonist cycle rather than a GnRH agonist cycle reduces significantly the risk of OHSS. During stimulation, the best predictor of severe OHSS is the number of follicles >10mm on the day of triggering final oocyte maturation, with the threshold at ≥16 follicles. When this occurs, final oocyte maturation can be induced with a GnRH agonist, reducing further the risk the syndrome. To perform a fresh embryo transfer, 1500 IU human Chorionic Gonadotropin (hCG) can be administered on the day of oocyte retrieval for the luteal support. However, with this procedure there are still some cases of OHSS. To overcome this, it is suggested to combine GnRH agonist triggering with a freeze-all embryos strategy and perform embryo replacement in subsequent frozen-thawed embryo transfer (FET) cycles. Different cryopreservation strategies are been performed according to the procedure of each fertility center, such as cryopreservation at 2 pronuclear (2PN), cleavage or blastocyst stage. The aim of this study is to determine the optimal strategy for the freeze-all cycles and particularly the optimal day for freezing, thawing and transferring the embryos. The hypothesis is that there will increased cumulative live birth rates per started cycle in blastocyst compared to cleavage stage FET cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients <40 years old
* Indication for In Vitro Fertilisation (IVF)/Intracytoplasmic sperm injection (ICSI)
* No more than 2 previous failed IVF/ICSI cycles
* Stimulation in GnRH antagonist cycle
* Presence of ≥16 follicles of >10mm on the day of triggering of final oocyte maturation
* GnRH agonist trigger (triptorelin 0.2mg)

Exclusion Criteria:

* Cycles with testicular sperm extraction
* Preimplantation genetic diagnosis
* Patients with uterine malformations
* Patients with infectious diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth | within one year of randomisation
  Cumulative live birth rate per oocyte retrieval

SECONDARY OUTCOMES:
Frozen thawed embryo transfer cycles needed to achieve live birth | within one year of randomisation
  Number of frozen thawed embryo transfer cycles needed to achieve live birth

IPD SHARING:
Plan to Share IPD: Undecided